CLINICAL TRIAL: NCT00437021
Title: Evaluation of IMVAMUNE® Smallpox Vaccine With Respect to Safety and Optimization of Immune Responses by Different Vaccination Regimens in Vaccinia-Naïve Adults
Brief Title: MVA Post-Event: Administration Timing and Boost Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-0012
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2010-03-08

CONDITIONS: Smallpox
Keywords: IMVAMUNE®; smallpox; vaccine
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group A (Experimental): Standard dose IMVAMUNE® vaccine or placebo on Days 0 and 7.
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo
- Group B (Experimental): Standard dose IMVAMUNE® vaccine or placebo on Days 0 and 28.
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo
- Group C (Active Comparator): Dryvax® vaccine or placebo on Day 0. This arm was discontinued from original protocol. Subjects already enrolled in this group will continue follow-up per protocol.
  Interventions: Biological: Live vaccinia virus vaccine; Other: Placebo
- Group D (Experimental): Standard dose IMVAMUNE® vaccine or placebo on Day 0 and Dryvax® vaccine or placebo on Day 7. This arm was discontinued from original protocol. Subjects already enrolled in this group will continue follow-up per protocol.
  Interventions: Biological: Live vaccinia virus vaccine; Biological: MVA Smallpox Vaccine; Other: Placebo
- Group E (Experimental): Dryvax® vaccine and standard dose IMVAMUNE® vaccine or 2 placebos on Day 0. This arm was discontinued from original protocol. Subjects already enrolled in this group will continue follow-up per protocol.
  Interventions: Biological: Live vaccinia virus vaccine; Biological: MVA Smallpox Vaccine; Other: Placebo
- Group F (Experimental): Standard dose IMVAMUNE® vaccine or placebo on Day 0.
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo

INTERVENTIONS:
Biological: Live vaccinia virus vaccine — Dryvax® Vaccinia Vaccine (~10^5 [plaque forming units (pfu)/dose] given via scarification, titer 10^8 pfu per mL after reconstitution).
  Arms: Group C; Group D; Group E
Biological: MVA Smallpox Vaccine — IMVAMUNE® Vaccinia Vaccine delivered by subcutaneous (SC) route at titer 1X10^8 Tissue Culture Infections Dose50 per 0.5 mL dose.
  Arms: Group A; Group B; Group D; Group E; Group F
Other: Placebo — 0.9 percent (weight/volume) sodium chloride injection, United States Pharmacopeia [Sterile Saline Placebo (SSP)].
  Arms: Group A; Group B; Group D; Group E; Group F
Other: Placebo — Physiologic normal saline for injection.
  Arms: Group C; Group D; Group E

SUMMARY:
The purpose of this study is to evaluate an investigational smallpox vaccine, called IMVAMUNE®, with respect to safety and immune (body's defense system) response. Participants will include healthy adults, age 18 or older born after 1971, who have not had smallpox vaccine before. Participants were originally assigned to 1 of 5 groups. In July 2007, a hold was placed on the Dryvax® groups and the study was modified. Participants, will be assigned by chance to one of 3 groups to be vaccinated twice with IMVAMUNE® vaccine or placebo (inactive substance) in Groups A and B, or to receive a single vaccination with IMVAMUNE® or placebo in Group F. Participants will complete a memory aid (diary) for 15 days following vaccination. Blood samples will be collected. Participants may participate for up to 425 days.

DETAILED DESCRIPTION:
The study will evaluate the IMVAMUNE® smallpox vaccine with respect to safety and optimization of immune responses by different vaccination regimens in vaccinia-naïve adults. Study participants must be age 18 and older and born after 1971. Originally, participants were planned to be randomly assigned to 1 of 5 groups to be immunized twice with IMVAMUNE® vaccine or placebo subcutaneously in Groups A and B, or Dryvax® or placebo by scarification in Group C or both IMVAMUNE® and Dryvax® or 2 placebos in Groups D and Group E. In July 2007, enrollment was halted at the request of Center for Biologics Evaluation and Research (CBER). At that time, enrollment included zero subjects in Group A, 2 subjects in Group B, 8 subjects in Group C, 6 subjects in Group D, and 4 subjects in Group E. CBER placed an official hold on the enrollment into the Groups that would administer Dryvax®, i.e., Groups C, D and E. Subjects previously enrolled into Groups C, D, and E will be followed according to the protocol. The protocol has been modified as follows. Participants will be randomly assigned to 1 of 3 groups to be immunized twice with IMVAMUNE® vaccine or placebo subcutaneously in Groups A and B, or to receive a single immunization with IMVAMUNE® or placebo subcutaneously in Group F. (NOTE: Group B will contain two additional participants that were enrolled prior to modification.) Group A will receive IMVAMUNE® vaccine or placebo on Days 0 and 7. Group B will receive IMVAMUNE® vaccine or placebo on Days 0 and 28. Group F will receive a single dose of IMVAMUNE® at Day 0. All participants will complete a memory aid for 15 days following each vaccination. Groups C, D, and E will have the appropriate reactogenicity information collected until the vaccination lesion, if present is well dried. Adverse events will be collected for 28 days after each vaccination. Specimens will be collected for immunologic assays at the noted clinic visits, as well as 1 year post last vaccination. Serious adverse events will be collected throughout the study period. The primary safety objective is to evaluate the safety of IMVAMUNE® given as a single dose, IMVAMUNE® given in a 2 dose prime-boost regimen at Day 0 and 7 or Day 0 and 28, IMVAMUNE® followed by a boost with Dryvax®, and IMVAMUNE® given simultaneously with Dryvax®. The primary immunogenicity objective is to determine if the Geometric Mean Titer (GMT) of neutralizing antibody [using Modified Vaccinia Ankara (MVA) as the target antigen] among subjects receiving a regimen of 2 doses of IMVAMUNE® (1×10^8, Days 0 and 7, Group A) is non-inferior to that among subjects receiving 2 doses of IMVAMUNE® (1×10^8, Days 0 and 28, Group B) at Day 14 following the 2nd dose. The secondary immunogenicity objective is to determine if the GMT, as assessed by enzyme linked immunosorbent assay (ELISA) (using MVA as the target antigen), among subjects receiving a regimen of 2 doses of IMVAMUNE® (1×10^8, Days 0 and 7, Group A) is non-inferior to that among subjects receiving 2 doses of IMVAMUNE® (1×10^8, Days 0 and 28, Group B) at Day 14 following the 2nd dose. The tertiary immunogenicity objective is to characterize the kinetics, magnitude, and duration of cellular and humoral immune responses to IMVAMUNE® alone or IMVAMUNE® as a prime followed by a boost with IMVAMUNE® or Dryvax®, or Dryvax® alone.

ELIGIBILITY:
Inclusion Criteria:

-At least 18 years of age and born after 1971 -Never received smallpox vaccination -Read, signed, and dated informed consent document -Available for follow-up for the planned duration of the study (one year after last immunization) -Acceptable medical history by screening evaluation and limited physical assessment -If the subject is female and of childbearing potential, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to vaccination -If the subject is female and of childbearing potential, she agrees to use acceptable contraception, and not become pregnant for the duration of the study a. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized b. Acceptable contraception methods are restricted to effective devices (e.g., Intrauterine Devices (IUD)s, NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, and abstinence from sexual intercourse with men (vaginal penetration by a penis, coitus) c. Women who are not sexually active must agree to use one of the acceptable contraception methods if they are of childbearing potential -Negative enzyme linked immunosorbent assay (ELISA) for human immunodeficiency virus (HIV) -Alanine aminotransferase (ALT) <1.25 times institutional upper limit of normal -Negative hepatitis B surface antigen and negative antibody to hepatitis C virus -Negative urine glucose and urine protein <1 plus by dipstick or urinalysis Adequate renal function defined as a serum creatinine equal to or less than the institutional upper limit of normal by gender; and urine protein <30 mg/dL or trace proteinuria (by urinalysis or dip stick). -Electrocardiogram (ECG) in absence of clinical significance (e.g., complete left or right bundle branch block, incomplete left bundle branch block or sustained ventricular arrythmia, or two premature ventricular contractions (PVC's) in a row, or sympathetic tonus (ST) elevation consistent with ischemia) -Complete blood count (CBC): Hemoglobin equal to or above the lower limit of institutional normal; White blood cells greater than or equal to 3200 /mm^3 and equal to or below the upper limit of institutional normal Platelets equal to or above the lower limit of institutional normal -Weight: greater than or equal to 110 pounds

Exclusion Criteria:

-History of immunodeficiency -Typical vaccinia scar -Known or suspected history of smallpox vaccination -Military service prior to 1991 or after January 2003 -Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease, diabetes mellitus, or moderate to severe kidney impairment -Malignancy not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site -Active autoimmune disease Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded. -History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor -Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp) -NOTE that this criterion applies only to subjects 20 years of age and older AND only if at least one of the following apply: a. have smoked a cigarette in the past month, and/or b. have hypertension (defined as systolic blood pressure >140 mm Hg) or are on antihypertensive medication, and/or c. have a family history of coronary heart disease in male first-degree relative (father or brother) <55 years of age or a female first-degree relative (mother or sister) <65 years of age. -Current use of immunosuppressive medication a. Corticosteroid nasal sprays are permissible b. Persons who are using a topical steroid can be enrolled after their therapy is completed c. Inhaled steroids for asthma are not permissible -Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol -Any history of illegal injection drug use -Receipt of inactivated vaccine 14 days prior to vaccination -Receipt of live attenuated vaccine within 30 days prior to vaccination -Use of experimental agent within 30 days prior to vaccination -Receipt of blood products or immunoglobulin within six months prior to vaccination -Donation of a unit of blood within 56 days prior to vaccination or for the duration of the study -Acute febrile illness (greater than or equal to 100.5 degrees F) on the day of vaccination -Pregnant or lactating women -Eczema of any degree or history of eczema -People with atopic dermatitis, chronic exfoliative skin disorders/conditions, current Varicella zoster, or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2×2 cm -Any condition that, in the opinion of the investigator, might interfere with study objectives -Known allergy to IMVAMUNE® vaccine -Known allergy to egg or aminoglycoside -Study personnel

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2007-04-16 (Actual); Primary Completion 2009-04-21 (Actual); Study Completion 2009-04-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Saint Louis University Center for Vaccine Development, St Louis, Missouri
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York
  - Duke Translational Medicine Institute - Clinical Vaccine Unit, Durham, North Carolina
  - Case Western Reserve University - John T. Carey Special Immunology Unit, Cleveland, Ohio
  - University of Texas Medical Branch - Pediatrics - Infectious Diseases and Immunology - Galveston, Galveston, Texas

REFERENCES:
- [Result] Frey SE, Winokur PL, Salata RA, El-Kamary SS, Turley CB, Walter EB Jr, Hay CM, Newman FK, Hill HR, Zhang Y, Chaplin P, Tary-Lehmann M, Belshe RB. Safety and immunogenicity of IMVAMUNE(R) smallpox vaccine using different strategies for a post event scenario. Vaccine. 2013 Jun 24;31(29):3025-33. doi: 10.1016/j.vaccine.2013.04.050. Epub 2013 May 9. PMID 23664987

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included adults aged greater than 18 years (and born after 1971) who met all inclusion/exclusion criteria. Participants were recruited from seven sites within the United States. The first participant was enrolled on April 16, 2007, and the last participant was enrolled on April 3, 2008.
Groups:
- Group A: Two Doses IMVAMUNE, Days 0, 7: Standard dose IMVAMUNE® vaccine on Days 0 and 7.
  IMVAMUNE®: IMVAMUNE® Vaccinia Vaccine delivered by subcutaneous (SC) route at titer 1X10^8 Tissue Culture Infections Dose50 per 0.5 mL dose.
- Group B: Two Doses IMVAMUNE, Days 0, 28: Standard dose IMVAMUNE® vaccine on Days 0 and 28.
  IMVAMUNE®: IMVAMUNE® Vaccinia Vaccine delivered by subcutaneous (SC) route at titer 1X10^8 Tissue Culture Infections Dose50 per 0.5 mL dose.
- Group C: One Dose Dryvax, Day 0: Dryvax® vaccine on Day 0. This arm was discontinued from original protocol. Participants already enrolled in this group continued follow-up per protocol.
  Dryvax®: Dryvax® Vaccinia Vaccine (~10^5 [plaque forming units (pfu)/dose] given via scarification, titer 10^8 pfu per mL after reconstitution).
- Group D: IMVAMUNE, Day 0 + Dryvax, Day 7: Standard dose IMVAMUNE® vaccine on Day 0 and Dryvax® vaccine on Day 7. This arm was discontinued from original protocol. Participants already enrolled in this group continued follow-up per protocol.
  Dryvax®: Dryvax® Vaccinia Vaccine (~10^5 [plaque forming units (pfu)/dose] given via scarification, titer 10^8 pfu per mL after reconstitution).
  IMVAMUNE®: IMVAMUNE® Vaccinia Vaccine delivered by subcutaneous (SC) route at titer 1X10^8 Tissue Culture Infections Dose50 per 0.5 mL dose.
- Group E: IMVAMUNE + Dryvax, Day 0: Dryvax® vaccine and standard dose IMVAMUNE® vaccine on Day 0. This arm was discontinued from original protocol. Participants already enrolled in this group continued follow-up per protocol.
  Dryvax®: Dryvax® Vaccinia Vaccine (~10^5 [plaque forming units (pfu)/dose] given via scarification, titer 10^8 pfu per mL after reconstitution).
  IMVAMUNE®: IMVAMUNE® Vaccinia Vaccine delivered by subcutaneous (SC) route at titer 1X10^8 Tissue Culture Infections Dose50 per 0.5 mL dose.
- Group F: IMVAMUNE, Day 0: Standard dose IMVAMUNE® vaccine on Day 0.
  IMVAMUNE®: IMVAMUNE® Vaccinia Vaccine delivered by subcutaneous (SC) route at titer 1X10^8 Tissue Culture Infections Dose50 per 0.5 mL dose.
- Placebo A: Placebo participants from Group A. Placebo administered corresponding to method for active drug administration in Group A.
  Placebo (subcutaneous): 0.9 percent (weight/volume) sodium chloride injection, United States Pharmacopeia [Sterile Saline Placebo (SSP)].
- Placebo B: Placebo participants from Group B. Placebo administered corresponding to method for active drug administration in Group B.
  Placebo (subcutaneous): 0.9 percent (weight/volume) sodium chloride injection, United States Pharmacopeia [Sterile Saline Placebo (SSP)].
- Placebo C: Placebo participants from Group C. Placebo administered corresponding to method for active drug administration in Group C.
  Placebo (scarification): Physiologic normal saline for injection.
- Placebo D: Placebo participants from Group D. Placebo administered corresponding to method for active drug administration in Group D.
  Placebo (subcutaneous): 0.9 percent (weight/volume) sodium chloride injection, United States Pharmacopeia [Sterile Saline Placebo (SSP)].
  Placebo (scarification): Physiologic normal saline for injection.
- Placebo E: Placebo participants from Group E. Placebo administered corresponding to method for active drug administration in Group E.
  Placebo (subcutaneous): 0.9 percent (weight/volume) sodium chloride injection, United States Pharmacopeia [Sterile Saline Placebo (SSP)].
  Placebo (scarification): Physiologic normal saline for injection.
- Placebo F: Placebo participants from Group F. Placebo administered corresponding to method for active drug administration in Group F.
  Placebo (subcutaneous): 0.9 percent (weight/volume) sodium chloride injection, United States Pharmacopeia [Sterile Saline Placebo (SSP)].
Period: Overall Study
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28 | Group C: One Dose Dryvax, Day 0 | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 | Group E: IMVAMUNE + Dryvax, Day 0 | Group F: IMVAMUNE, Day 0 | Placebo A | Placebo B | Placebo C | Placebo D | Placebo E | Placebo F
Started | 61 | 66 | 8 | 5 | 2 | 63 | 6 | 5 | 0 | 1 | 2 | 7
Completed | 59 | 62 | 8 | 5 | 2 | 61 | 5 | 4 | 0 | 1 | 2 | 7
Not Completed | 2 | 4 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were analyzed according to the treatment group they were randomized to.
Groups:
- Group A: Two Doses IMVAMUNE, Days 0, 7: Standard dose IMVAMUNE® vaccine on Days 0 and 7.
- Group B: Two Doses IMVAMUNE, Days 0, 28: Standard dose IMVAMUNE® vaccine on Days 0 and 28.
- Group C: One Dose Dryvax, Day 0: Dryvax® vaccine on Day 0. This arm was discontinued from original protocol. Participants already enrolled in this group continued follow-up per protocol.
- Group D: IMVAMUNE, Day 0 + Dryvax, Day 7: Standard dose IMVAMUNE® vaccine on Day 0 and Dryvax® vaccine on Day 7. This arm was discontinued from original protocol. Participants already enrolled in this group continued follow-up per protocol.
- Group E: IMVAMUNE + Dryvax, Day 0: Dryvax® vaccine and standard dose IMVAMUNE® vaccine on Day 0. This arm was discontinued from original protocol. Participants already enrolled in this group continued follow-up per protocol.
- Group F: IMVAMUNE, Day 0: Standard dose IMVAMUNE® vaccine on Day 0.
- Placebo A: Placebo participants from Group A. Placebo administered corresponding to method for active drug administration in Group A.
- Placebo B: Placebo participants from Group B. Placebo administered corresponding to method for active drug administration in Group B.
- Placebo D: Placebo participants from Group D. Placebo administered corresponding to method for active drug administration in Group D.
- Placebo E: Placebo participants from Group E. Placebo administered corresponding to method for active drug administration in Group E.
- Placebo F: Placebo participants from Group F. Placebo administered corresponding to method for active drug administration in Group F.
- Total: Total of all reporting groups
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28 | Group C: One Dose Dryvax, Day 0 | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 | Group E: IMVAMUNE + Dryvax, Day 0 | Group F: IMVAMUNE, Day 0 | Placebo A | Placebo B | Placebo D | Placebo E | Placebo F | Total
Number analyzed (Participants) | 61 | 66 | 8 | 5 | 2 | 63 | 6 | 5 | 1 | 2 | 7 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (4.6) | 25.0 (3.9) | 26.5 (4.3) | 26.4 (5.1) | 31.0 (4.2) | 24.3 (3.9) | 25.2 (3.5) | 21.4 (2.3) | 24.0 (NA) — Not estimable because only one participant was enrolled and randomized to this treatment group. | 20.5 (0.7) | 27.9 (4.8) | 24.8 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 36 | 1 | 2 | 1 | 32 | 3 | 0 | 0 | 0 | 5 | 105
  Male | 36 | 30 | 7 | 3 | 1 | 31 | 3 | 5 | 1 | 2 | 2 | 121
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 9
  Not Hispanic or Latino | 59 | 63 | 8 | 5 | 2 | 60 | 5 | 5 | 1 | 2 | 7 | 217
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 0 | 1 | 0 | 6 | 0 | 0 | 0 | 0 | 1 | 16
  White | 52 | 56 | 8 | 4 | 2 | 54 | 6 | 4 | 1 | 2 | 6 | 195
  More than one race | 4 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 8
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Bavarian Nordic's (BN) Plaque Reduction Neutralizing Antibody Titer (PRNT) Assay in Groups A and B
Description: Geometric mean of titers collected 14 days after the second vaccination.
Time Frame: Day 14 after the second vaccination
Population: The analysis population includes all participants who received two doses of study vaccine and contributed both pre- and post-vaccination blood samples for testing for which valid results were reported. Participants were analyzed "as treated" according to the study product they received.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28
Number analyzed (Participants) | 59 | 63
titer | 10.8 [9.0 to 12.9] | 30.2 [22.1 to 41.1]
Statistical Analysis 1: Comparison: Group A: Two Doses IMVAMUNE, Days 0, 7 vs Group B: Two Doses IMVAMUNE, Days 0, 28; Null hypothesis: The mean difference in log2 transformed titers between Group B and Group A >= 1; Test type: Non-Inferiority — The non-inferiority margin is 1. Non-inferiority of Group A is concluded if the upper limit of the 95% confidence interval for the mean difference in the log2 transformed peak titers between groups is less than 1; Mean Difference (Final Values) = 1.48, 95% CI 2-sided [0.97 to 1.99] — Estimate and corresponding 95% confidence interval are calculated on the log2 scale

2. Primary Outcome: GMT of Saint Louis University's (SLU) PRNT Assay in Group A and Group B
Description: Geometric mean of titers collected 14 days after the second vaccination.
Time Frame: Day 14 after the second vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28
Number analyzed (Participants) | 59 | 63
titer | 27.4 [19.1 to 39.3] | 212.2 [146.6 to 307.2]
Statistical Analysis 1: Comparison: Group A: Two Doses IMVAMUNE, Days 0, 7 vs Group B: Two Doses IMVAMUNE, Days 0, 28; Null hypothesis: The mean difference in log2 transformed titers between Group B and Group A >= 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.895, 95% CI 2-sided [2.22 to 3.69] — Estimate and corresponding 95% confidence interval are calculated on the log2 scale

3. Primary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: The number of participants who experienced at least one SAE throughout the course of the study. A SAE is defined as an AE meeting one of the following conditions:
  * Death during the study period (from first vaccine until end of surveillance period)
  * Life-threatening (defined as a participant at immediate risk of death at the time of the event)
  * Requires inpatient hospitalization or prolongation of existing hospitalization during the period of protocol-defined surveillance
  * Results in a congenital anomaly or birth defect
  * Results in a persistent or significant disability/incapacity
  * Severe adverse event associated with study product
Time Frame: Day 0 after first vaccination to study completion through Day 365 after last vaccination
Population: The safety population includes all participants who received one dose of vaccine. Participants were analyzed "as treated" according to the study product they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28 | Group C: One Dose Dryvax, Day 0 | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 | Group E: IMVAMUNE + Dryvax, Day 0 | Group F: IMVAMUNE, Day 0 | Placebo A | Placebo B | Placebo D | Placebo E | Placebo F
Number analyzed (Participants) | 61 | 67 | 8 | 5 | 2 | 63 | 6 | 4 | 1 | 2 | 7
Participants | 1 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Frequency of Non-Serious AEs
Description: The number of participants who experienced at least one unsolicited non-serious AE of any severity from Day 0 after the first vaccination to 28 days after the last vaccination.
Time Frame: Day 0 after first vaccination through Day 28 after last vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28 | Group C: One Dose Dryvax, Day 0 | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 | Group E: IMVAMUNE + Dryvax, Day 0 | Group F: IMVAMUNE, Day 0 | Placebo A | Placebo B | Placebo D | Placebo E | Placebo F
Number analyzed (Participants) | 61 | 67 | 8 | 5 | 2 | 63 | 6 | 4 | 1 | 2 | 7
Participants | 32 | 43 | 4 | 1 | 0 | 26 | 4 | 2 | 0 | 0 | 5

5. Primary Outcome: Frequency of Local Solicited Reactogenicity AEs for Groups A, B, and D and Placebo A, B, and D
Description: Local solicited reactogenicity AEs were collected daily for 15 days post each vaccination using a memory aid. Local events include pain at vaccination site, itchiness at vaccination site, rash at vaccination site underarm pain, underarm swelling, erythema, and induration. Erythema and induration at the vaccination site were measured in millimeters; the remaining events were graded on a subjective scale of Grade 0 (None), Grade 1 (Mild), Grade 2 (Moderate), and Grade 3 (Severe).
Time Frame: Day 0 through Day 15 after first vaccination; Day 0 through Day 15 after second vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28 | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 | Placebo A | Placebo B | Placebo D
Number analyzed (Participants) | 61 | 67 | 5 | 6 | 4 | 1
Participants
  Post First Vaccination | 47 | 50 | 4 | 1 | 2 | 0
  Post Second Vaccination: number analyzed (Participants) | 59 | 64 | 3 | 5 | 3 | 1
  Post Second Vaccination | 51 | 53 | 3 | 0 | 0 | 1

6. Primary Outcome: Frequency of Local Solicited Reactogenicity AEs for Groups C and F and Placebo F
Description: Local solicited reactogenicity AEs were collected daily for 15 days post vaccination using a memory aid. Local events include pain at vaccination site, itchiness at vaccination site, rash at vaccination site underarm pain, underarm swelling, erythema, and induration. Erythema and induration at the vaccination site were measured in millimeters; the remaining events were graded on a subjective scale of Grade 0 (None), Grade 1 (Mild), Grade 2 (Moderate), and Grade 3 (Severe).
Time Frame: Day 0 through Day 15 after first vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group C: One Dose Dryvax, Day 0 | Group F: IMVAMUNE, Day 0 | Placebo F
Number analyzed (Participants) | 8 | 63 | 7
Participants | 8 | 50 | 1

7. Primary Outcome: Frequency of Local Solicited Reactogenicity AEs for Group E and Placebo E
Description: Local solicited reactogenicity AEs were collected daily for 15 days post vaccination using a memory aid. Results are reported by vaccination site (MVA Vaccination or Dryvax Vaccination). Local events included pain at vaccination site, itchiness at vaccination site, rash at vaccination site underarm pain, underarm swelling, erythema, and induration. Erythema and induration at the vaccination site were measured in millimeters; the remaining events were graded on a subjective scale of Grade 0 (None), Grade 1 (Mild), Grade 2 (Moderate), and Grade 3 (Severe).
Time Frame: Day 0 through Day 15 after first vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group E: IMVAMUNE + Dryvax, Day 0 | Placebo E
Number analyzed (Participants) | 2 | 2
Participants
  MVA Vaccination | 1 | 0
  Dryvax Vaccination | 2 | 2

8. Primary Outcome: Frequency of Systemic Solicited Reactogenicity AEs for Groups A, B, and D and Placebo A, B, and D
Description: Systemic solicited reactogenicity AEs were collected daily for 15 days post each vaccination using a memory aid. Systemic events included muscle aches, chills, headache, nausea, feeling tired, change in appetite, joint pain, and elevated oral temperature. Events were graded on a subjective scale of Grade 0 (None), Grade 1 (Mild), Grade 2 (Moderate), and Grade 3 (Severe).
Time Frame: Day 0 through Day 15 after first vaccination; Day 0 through Day 15 after second vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28 | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 | Placebo A | Placebo B | Placebo D
Number analyzed (Participants) | 61 | 67 | 5 | 6 | 4 | 1
Participants
  Post First Vaccination | 31 | 41 | 2 | 4 | 3 | 0
  Post Second Vaccination: number analyzed (Participants) | 59 | 64 | 3 | 5 | 3 | 1
  Post Second Vaccination | 29 | 23 | 3 | 2 | 3 | 0

9. Primary Outcome: Frequency of Systemic Solicited Reactogenicity AEs for Groups C, E, and F and Placebo E and F
Description: Systemic solicited reactogenicity AEs were collected daily for 15 days post vaccination using a memory aid. Systemic events included muscle aches, chills, headache, nausea, feeling tired, change in appetite, joint pain, and elevated oral temperature. Events were graded on a subjective scale of Grade 0 (None), Grade 1 (Mild), Grade 2 (Moderate), and Grade 3 (Severe).
Time Frame: Day 0 through Day 15 after first vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group C: One Dose Dryvax, Day 0 | Group E: IMVAMUNE + Dryvax, Day 0 | Group F: IMVAMUNE, Day 0 | Placebo E | Placebo F
Number analyzed (Participants) | 8 | 2 | 63 | 2 | 7
Participants | 5 | 2 | 33 | 1 | 3

10. Secondary Outcome: GMT of BN Enzyme Linked Immunosorbent Assay (ELISA) in Groups A and B
Description: Geometric mean of titers collected 14 days after the second vaccination.
Time Frame: Day 14 after the second vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28
Number analyzed (Participants) | 59 | 63
titer | 108.7 [87.7 to 134.8] | 501.7 [364.1 to 691.3]
Statistical Analysis 1: Comparison: Group A: Two Doses IMVAMUNE, Days 0, 7 vs Group B: Two Doses IMVAMUNE, Days 0, 28; Null hypothesis: The mean difference in log2 transformed titers between Group B and Group A >= 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.21, 95% CI 2-sided [1.65 to 2.76] — Estimate and corresponding 95% confidence interval are calculated on the log2 scale

11. Secondary Outcome: GMT of SLU ELISA in Groups A and B
Description: Geometric mean of titers collected 14 days after the second vaccination.
Time Frame: Day 14 after the second vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28
Number analyzed (Participants) | 59 | 63
titer | 60.5 [51.0 to 71.7] | 510.9 [373.0 to 699.7]
Statistical Analysis 1: Comparison: Group A: Two Doses IMVAMUNE, Days 0, 7 vs Group B: Two Doses IMVAMUNE, Days 0, 28; Null hypothesis: The mean difference in log2 transformed titers between Group B and Group A >= 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 3.08, 95% CI 2-sided [2.57 to 3.59] — Estimate and corresponding 95% confidence interval are calculated on the log2 scale

ADVERSE EVENTS:
Time Frame: AEs collected include solicited AEs, unsolicited AEs, and SAEs. Solicited AEs were collected daily for 15 days post each vaccination. Unsolicited AEs were collected from the first vaccination through 28 days after the last vaccination. SAEs were collected from the first vaccination to study completion (Day 365 after the last vaccination).
Description: Participants were analyzed "as treated" according to the study product they received. One participant enrolled in Group B was randomized to Placebo B but was actually administered two doses IMVAMUNE on Days 0 and 28. For AE results, this participant is counted among those at risk in Group B: Two Doses IMVAMUNE, Days 0, 28.
Arm/Group | Group A: Two Doses IMVAMUNE, Days 0, 7 | Group B: Two Doses IMVAMUNE, Days 0, 28 | Group C: One Dose Dryvax, Day 0 | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 | Group E: IMVAMUNE + Dryvax, Day 0 | Group F: IMVAMUNE, Day 0 | Placebo A | Placebo B | Placebo D | Placebo E | Placebo F
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/67 | 0/8 | 0/5 | 0/2 | 0/63 | 0/6 | 0/4 | 0/1 | 0/2 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/61 | 2/67 | 0/8 | 0/5 | 0/2 | 3/63 | 0/6 | 0/4 | 0/1 | 0/2 | 0/7
Other Adverse Events (participants affected / at risk) | 57/61 | 66/67 | 8/8 | 5/5 | 2/2 | 58/63 | 6/6 | 4/4 | 1/1 | 2/2 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Two Doses IMVAMUNE, Days 0, 7 (N=61) | Group B: Two Doses IMVAMUNE, Days 0, 28 (N=67) | Group C: One Dose Dryvax, Day 0 (N=8) | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 (N=5) | Group E: IMVAMUNE + Dryvax, Day 0 (N=2) | Group F: IMVAMUNE, Day 0 (N=63) | Placebo A (N=6) | Placebo B (N=4) | Placebo D (N=1) | Placebo E (N=2) | Placebo F (N=7)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complicated migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteral disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cosmetic surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Two Doses IMVAMUNE, Days 0, 7 (N=61) | Group B: Two Doses IMVAMUNE, Days 0, 28 (N=67) | Group C: One Dose Dryvax, Day 0 (N=8) | Group D: IMVAMUNE, Day 0 + Dryvax, Day 7 (N=5) | Group E: IMVAMUNE + Dryvax, Day 0 (N=2) | Group F: IMVAMUNE, Day 0 (N=63) | Placebo A (N=6) | Placebo B (N=4) | Placebo D (N=1) | Placebo E (N=2) | Placebo F (N=7)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site dermatitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 7 (8) | 9 (9) | 5 (5) | 0 (0) | 1 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 5 (5) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 23 (29) | 24 (29) | 4 (4) | 4 (4) | 2 (2) | 23 (23) | 2 (3) | 4 (5) | 0 (0) | 1 (1) | 1 (1)
Injection site rash (General disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Underarm swelling (General disorders) | 5 (6) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site erythema (General disorders) | 34 (50) | 39 (53) | 8 (8) | 3 (3) | 2 (3) | 23 (23) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vaccination site pain (General disorders) | 52 (85) | 59 (94) | 5 (5) | 4 (5) | 1 (1) | 45 (45) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Vaccination site pruritus (General disorders) | 18 (21) | 15 (20) | 7 (7) | 2 (2) | 2 (3) | 11 (11) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vaccination site swelling (General disorders) | 29 (39) | 30 (42) | 7 (7) | 3 (3) | 2 (2) | 14 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 8 (8) | 8 (9) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 5 (5) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (25) | 19 (24) | 4 (4) | 0 (0) | 2 (2) | 13 (13) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 21 (24) | 30 (39) | 2 (2) | 1 (2) | 2 (2) | 24 (24) | 2 (3) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 10 (11) | 9 (13) | 2 (2) | 0 (0) | 1 (1) | 8 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less